CLINICAL TRIAL: NCT00424840
Title: Phase I/II Study to Evaluate the Efficacy and Safety of Combination Chemotherapy With Carboplatin, Bortezomib and Bevacizumab as First Line Therapy in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Phase I/II Study to Evaluate the Efficacy and Safety of a Combination Chemotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, William Walsh, Study Principle Investigator, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UM200601
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Lung Cancer
Keywords: lung cancer, Carboplatin, bortezomib, Bevacizumab
MeSH Terms: conditions — Lung Neoplasms | interventions — Bortezomib; Carboplatin; Bevacizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Bortezomib 1.3 mg/m2 (Experimental): Level 1 of Bortezomib Dose Escalation in combination with Carboplatin AUC6, Bevacizumab 15 mg/kg and Taxotere 70 + G-CSF
  Interventions: Drug: Bortezomib 1.3 mg/m2; Drug: Carboplatin AUC 6; Drug: Bevacizumab; Drug: Taxotere
- Bortezomib 1.6 mg/m2 (Experimental): Level 2 of Bortezomib Dose Escalation in combination with Carboplatin AUC6, Bevacizumab 15 mg/kg and Taxotere 70 + G-CSF
  Interventions: Drug: Bortezomib 1.6 mg/m2; Drug: Carboplatin AUC 6; Drug: Bevacizumab; Drug: Taxotere
- Bortezomib 1.8 mg/m2 (Experimental): Level 3 of Bortezomib Dose Escalation in combination with Carboplatin AUC6, Bevacizumab 15 mg/kg and Taxotere 70 + G-CSF
  Interventions: Drug: Bortezomib 1.8 mg/m2; Drug: Carboplatin AUC 6; Drug: Bevacizumab; Drug: Taxotere

INTERVENTIONS:
Drug: Bortezomib 1.3 mg/m2 — Level I (every 21 day cycle, D8), 1.3 mg/m2:
  Day 1: bevacizumab 15 mg/kg ,carboplatin Area Under the Curve (AUC 6) 900mg, bortezomib 1.3 mg/m2 Day 8 : bortezomib 1.3 mg/m2
  Level II (every 21 day cycle):
  Day 1: bevacizumab 15 mg/kg, carboplatin Area Under the Curve (AUC 6) 900mg, bortezomib 1.6 mg/m2 Day 8 : bortezomib 1.6 mg/m2
  Level III(every 21 day cycle):
  Day 1: bevacizumab 15 mg/kg, carboplatin Area Under the Curve (AUC 6) 900mg, bortezomib 1.8 mg/m2 Day 8 : bortezomib 1.8 mg/m2
  Other Names: Velcade
  Arms: Bortezomib 1.3 mg/m2
Drug: Bortezomib 1.6 mg/m2 — Level II (every 21 day cycle, D8), 1.6 mg/m2
  Other Names: Velcade
  Arms: Bortezomib 1.6 mg/m2
Drug: Bortezomib 1.8 mg/m2 — Level III (every 21 day cycle, D8) 1.8 mg/m2
  Other Names: Velcade
  Arms: Bortezomib 1.8 mg/m2
Drug: Carboplatin AUC 6 — Carboplatin AUC6
  Other Names: Carboplatin
Drug: Bevacizumab — Bevacizumab 15 mg/kg
Drug: Taxotere — Taxotere 70 + G-CSF

SUMMARY:
A pilot trial of combination of bortezomib, bevacizumab and carboplatin as first line therapy in patients with metastatic Non-Small Cell Lung Cancer (NSCLC). Phase I and II study of this combination in first line setting will be conducted in order to properly estimate the efficacy and safety of this regimen. This will form the basis for future studies comparing this combination to what is now considered standard regimen for first line therapy in patients with NSCLC, carboplatin, paclitaxel and bevacizumab.

DETAILED DESCRIPTION:
Study design and methodology The study will have two phases.

The phase I will use traditional dose escalation model (3-6 patient per dose level) to determine the maximum tolerated dose (MTD).

*[In phase II, either level III or (MTD) will be used in the same every 21 day cycle to evaluate the efficacy and safety of the regimen in first line treatment of advanced NSCLC]* not conducted.

Treatments administered

In phase I, three dose levels of weekly bortezomib will be studied in conjunction with fixed dose carboplatin and bevacizumab on a 21 day cycle to define the maximum tolerated dose (MTD).

A maximum of six cycles will be administered. Patients with complete response, partial response or stable disease after six cycles will be allowed to continue on single agent bevacizumab every 3 weeks as maintenance therapy until disease progression.

If no dose limiting toxicity (DLT) is observed in 3 patients during the first cycle, the next dose level will be accrued. If 1 DLT is observed, 3 additional patients will be accrued to the dose level. If no additional DLTs are observed, the next dose level will be accrued. However, if 2 or more DLTs are observed in a given dose level, MTD will be defined. MTD will be defined as the dose below which ≥2 DLTs were observed.

The following three levels will be studied:

Level I (every 21 day cycle): D1: carboplatin AUC 6, bevacizumab 15 mg/kg, bortezomib 1.3 mg/m2 D8 : bortezomib 1.3 mg/m2

Level II (every 21 day cycle): D1: carboplatin AUC 6, bevacizumab 15 mg/kg, bortezomib 1.6 mg/m2 D8 : bortezomib 1.6 mg/m2

Level III(every 21 day cycle):D1: carboplatin AUC 6, bevacizumab 15 mg/kg, bortezomib 1.8 mg/m2 D8 : bortezomib 1.8 mg/m2

If 2 or more DLT are observed in Level 1, level -1 will be accrued.

Level -1: (every 21 day cycle): D1: carboplatin AUC 6, bevacizumab 15 mg/kg, bortezomib 1 mg/m2 D8: bortezomib 1 mg/m2

*[In phase II, either level III or the MTD dose level will be used in the same every 21 day cycle to evaluate the efficacy and safety of the regimen in first line treatment of advanced NSCLC.

Efficacy data collected

The following evaluations will be conducted to assess the efficacy of the combination:

* response rate by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* disease free and overall survival, time to progress (TTP) and duration of response Safety data collected

The following evaluations will be conducted to assess the safety of the combination chemotherapy:

• toxicity based on National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 3.0]* Not conducted

Statistical procedures

In phase I portion, 9-18 patients will be enrolled. The patients treated at recommended dose level for phase II will also be eligible for response evaluation as part of phase II.

*[The primary objective of the phase II study is to estimate the efficacy and safety of the combination therapy with carboplatin, bortezomib and bevacizumab as the first line therapy in patients with advanced NSCLC. The primary endpoints are response rate and progression-free survival (PFS).

(NOT CONDUCTED) In phase II portion, the optimal two-stage design for phase II clinical trials described by Simon et al. will be utilized.

Overall survival, progression free survival and time to progression will be estimated using Kaplan-Meier methods. Time to progression, progression free survival and survival will be calculated from the date of study entry.]* (Phase II not conducted.)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed SCLC (adeno- and large cell, anaplastic carcinoma and broncho-alveolar-carcinoma). Patients with squamous-cell histology are eligible with extra thoracic or peripheral lung lesions only.
* Sputum cytology alone not acceptable evidence of cell type. Cytologic specimens obtained by brushing, washings, or needle aspiration of defined lesions will be acceptable. Mixed tumors will be categorized by the predominant cell type unless a small cell anaplastic elements are present, in which case the patient is ineligible.
* Stage III B because of pleural effusion or Stage IV disease
* Measurable disease.
* Age: 18 years or older
* No history of thrombotic, hemorrhagic, or coagulopathy disorders
* international normalized ratio (INR<1.5) and a prothrombin time (PTT) no greater than normal limits of normal within 1 week prior to registration. NB: subjects with lung cancer placed on anticoagulant therapy for a thrombotic event are not eligible for this study.
* No gross hemoptysis (defined as bright red blood of ½ teaspoon or more)
* No central nervous system (CNS) or brain metastasis
* Laboratory Criteria (completed <2 weeks before enrollment):

  * Hematologic: white blood cell (WBC) > 3500/mm3 or absolute neutrophil count (ANC) > 1500/mm3 and platelet count > 100 000/ mm3;
  * Hepatic: Total bilirubin < 1.5 mg/dl
  * Renal: Creatinine < 1.5 mg/dl. or calculated
  * Creatinine clearance > 45 ml/min (NB: Urine protein:creatinine ratio in exclusion criteria)
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Be free of active infection.
* Be available for active follow up.
* No prior chemotherapy for metastatic disease.
* Be disease free for > 5 years if they had a prior second malignancy other than treated basal cell carcinoma or squamous cell skin cancer, or carcinoma in situ of the cervix.
* Female subject post-menopausal; surgically sterilized or willing to use an acceptable method of birth control for the duration of the study. Male subject agrees to use an acceptable method for contraception for the duration of the study.

Exclusion Criteria:

* CNS or brain metastasis
* Patient has = or greater Grade 2 peripheral neuropathy within 14 days before enrollment.
* Known previous sensitivity reactions with boron, or mannitol,
* Patients with known HIV positivity
* Myocardial infarction within 6 months prior to enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Blood pressure of >150/100 mmHG
* History of myocardial infarction or stroke within 6 months
* Clinically significant peripheral vascular disease
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedure such as fine needle aspirations or core biopsies within 7 days prior to day 0
* Urine protein: Creatinine ratio > 1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Lung carcinoma or any histology in close proximity to a major vessel or cavitation
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs with 14 days before enrollment or is expected to participate in an experiment drug study during this study treatment.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Walsh, MD, Principal Investigator — University of MassachusettsMedical School
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Sandler A, Gray R, Perry MC, Brahmer J, Schiller JH, Dowlati A, Lilenbaum R, Johnson DH. Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung cancer. N Engl J Med. 2006 Dec 14;355(24):2542-50. doi: 10.1056/NEJMoa061884. PMID 17167137

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Treatment q21 day cycle, maximum of 6 cycles. Patients with CR, PR, SD continued on single agent bevacizumab 15 mb/kg q 3 weeks.
Groups:
- Dose Level 1: 1.3 mg/m^2 Bortezomib: Level 1 participants were given 1.3 mg/m^2 Bortezomib with Carboplatin AUC6, bevacizumab 15 mg/kg
- Dose Level II: 1.6 mg/m^2: Participants were given1.6 mg/m^2 Bortezomib with Carboplatin AUC6, bevacizumab 15 mg/kg
- Dose Level III: 1.8 mg/m^2: 1.8 mg/m^2 Bortezomib with Carboplatin AUC6, bevacizumab 15 mg/kg
Period: Overall Study
Arm/Group | Dose Level 1: 1.3 mg/m^2 Bortezomib | Dose Level II: 1.6 mg/m^2 | Dose Level III: 1.8 mg/m^2
Started | 3 | 4 | 5
Completed | 3 | 4 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Dose Level 1, 2 and 3: 1.3 mg/m^2 Bortezomib", "1.6 mg/m^2 Bortezomib", and "1.8 mg/m^2 Bortezomib
  In phase I, three dose levels of weekly bortezomib will be studied in conjunction with fixed dose carboplatin and bevacizumab on a 21 day cycle to define the maximum tolerated dose (MTD).
Arm/Group | Phase I: Dose Level 1, 2 and 3
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 63 [49 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Require Dose Delay/Reduction in Dose of Bortezomibin the First Cycle
Description: Dose limiting toxicity at Level 1,2 and 3: Number of subjects who required dose delay/reduction in dose of bortezomib in the first cycle of treatment. DLT defined by any of the following during first cycle: (1) GR4 neutropenia or thrombocytopenia, (2) Greater than GR3 non-hematological toxicity except alopecia or inadequately treated nausea or vomiting or (3) neurosensory toxicity of GR2 with pain or any neurotoxicity greater than GR2.
Time Frame: up to 21 days for each dosing cycle
Measure: Number; unit: participants
Groups:
- Phase I: Dose Level 1: 1.3 mg/m^2 Bortezomib
- Phase 1 Dose Level II:: 1.6 mg/m^2 Bortezomib
- Phase I Dose Level III: 1.8 mg/m^2 Bortezomib
Arm/Group | Phase I: Dose Level 1 | Phase 1 Dose Level II: | Phase I Dose Level III
Number analyzed (Participants) | 3 | 4 | 5
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: From date of first dose to date of death or up to 2 years, whichever came first Adverse event data by separate arms not available
Groups:
- Phase I: Bevacizumab, Carboplatin, Bortezomib: In phase I, three dose levels of weekly bortezomib will be studied in conjunction with fixed dose carboplatin and bevacizumab on a 21 day cycle to define the maximum tolerated dose (MTD).
  Bevacizumab will be administered first followed by carboplatin followed by bortezomib
Arm/Group | Phase I: Bevacizumab, Carboplatin, Bortezomib
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 7/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Bevacizumab, Carboplatin, Bortezomib (N=12)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4)
Hyponatremia (Blood and lymphatic system disorders) | 5 (5)
Peripheral Neuropathy (Vascular disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
The study was closed prematurely because of poor accrual prior to initiation of Phase 2, and is underpowered to definitely estimated the response rate and progression free survival.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No